CLINICAL TRIAL: NCT00895193
Title: Alternative Options to Minimize Niacin-Induced Flushing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Moriarty, MD, FACP, FACC (Other)
Responsible Party: Sponsor-Investigator, Patrick Moriarty, MD, FACP, FACC, Director, Clinical Pharmacology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11627
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Hypercholesterolemia; Flushing
Keywords: Niacin; Hypercholesterolemia; Flushing
MeSH Terms: conditions — Hypercholesterolemia; Flushing | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Apple-pectin 2000mg (Active Comparator): Participant receives Apple pectin 2000mg 30 minutes prior to a one-time 1000mg dose of extended-release niacin.
  Interventions: Other: Apple pectin
- Regular Non-enteric coated aspirin 325mg (Active Comparator): Participant receives aspirin 325 mg 30 minutes prior to a one-time 1000mg dose of extended-release niacin.
  Interventions: Drug: Aspirin 325 mg
- Apple pectin + aspirin (Active Comparator): Participant receives apple pectin 2000mg and aspirin 325 mg 30 minutes prior to a one-time 1000mg dose of extended-release niacin.
  Interventions: Other: Apple pectin; Drug: Aspirin 325 mg
- Placebo Comparator (Placebo Comparator): Participant receives placebo 30 minutes prior to a one-time 1000mg dose of extended-release niacin.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Apple pectin — Apple pectin 2000mg
  Arms: Apple pectin + aspirin; Apple-pectin 2000mg
Drug: Aspirin 325 mg — Aspirin 325 mg
  Arms: Apple pectin + aspirin; Regular Non-enteric coated aspirin 325mg
Other: Placebo — Placebo
  Arms: Placebo Comparator

SUMMARY:
Niacin (Vitamin B3) is known to effectively and safely treat hypercholesterolemia. However, use of niacin is limited due to incidents of flushing which limits its acceptability. Some information suggests that applesauce can reduce the incidence and severity of flushing. The apple pectin in particular is thought to be the ingredient that affects this reaction. To determine if the apple pectin does affect flushing from niacin, the investigators will study the affects of isolated apple pectin in pill form. The investigators plan on recruiting 100 patients, and giving them 1000 mg of Niacin to induce flushing. Patients will be divided into 4 treatment groups and receive either pectin, aspirin, a combination of both, or placebo. Incidents and severity of flushing will be monitored for up to 6 hours post Niacin ingestion.

ELIGIBILITY:
Inclusion Criteria:

* An adult between 21 and 70 years of age.
* Male or female (If female must be postmenopausal for at least 1 year, surgically sterile or using an effective form of contraception).
* Able to speak and read English.
* Willing to comply with study specific instructions, and complete all study procedures according to protocol.
* Able to understand study rationale and sign informed consent.

Exclusion Criteria:

* Females of child-bearing potential not using acceptable method of contraception and perimenopausal females.
* History of gout
* History of diabetes mellitus
* History of coronary heart disease
* History of, or currently experiencing, renal disease including, but not limited to, renal insufficiency, nephrolithiasis or chronic renal failure.
* History of, or currently experiencing, major chronic gastrointestinal condition including gallbladder disease, liver disease and peptic ulcer disease
* Known sensitivity to niacin, Aspirin or nonsteroidal anti-inflammatory agents (NSAIDs)
* History of migraine or cluster headaches
* Currently using antihistamines, aspirin or NSAIDS on a consistent basis
* Presence or history of any medical or psychosocial condition that, in the opinion of the investigator, would limit the patient's successful participation or would compromise the patient's safe participation.
* Lab abnormalities at screening, including but not limited to elevated liver enzymes or blood sugar levels that might indicate additional risk to the patient's continued participation.
* Currently taking medication that might be contraindicated with the study drug or Niacin or study procedures (including Niacin, lipid-lowering drugs, chronic aspirin or laxative use).
* Clinically significant finding from physical exam that would affect the patient's safe participation or completion of the study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Moriarty, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial screening occurred over the telephone. Subjects that met preliminary study criteria were scheduled for a screening visit. Recruitment was conducted at the University of Kansas Medical Center.
Period: Overall Study
Arm/Group | Apple-pectin 2000mg | Regular Non-enteric Coated Aspirin 325mg | Apple Pectin + Aspirin | Placebo Comparator
Started | 25 | 25 | 25 | 25
Completed | 25 | 25 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apple-pectin 2000mg | Regular Non-enteric Coated Aspirin 325mg | Apple Pectin + Aspirin | Placebo Comparator | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11.5) | 40 (13.3) | 40 (12.3) | 38 (12.7) | 38.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 11 | 11 | 45
  Male | 14 | 13 | 14 | 14 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 9 | 5 | 5 | 23
  White | 16 | 15 | 20 | 20 | 71
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 25 | 100
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26 (5.5) | 27 (6.2) | 26 (5.3) | 26 (5.0) | 26.4 (5.4)
Waist Circumference [Mean (Standard Deviation); unit: inches] | 35 (6.1) | 36 (6.3) | 34 (5.0) | 35 (5.3) | 35 (5.65)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Flushing
Description: Flushing assessment performed hourly for 6 hours after niacin administration. Incidence of flushing based on if the participant experience any niacin-induced flushing during the 6 hour period after dosing. Represents # of participants that experienced event.
Time Frame: Hourly for 6 hours on day of dosing
Population: This was a single-site, randomized trial, 4-arm parallel design trial. Each arm consisted of 25 randomized participants. All participants completed the study.
Measure: Number; unit: participants
Arm/Group | Apple-pectin 2000mg | Regular Non-enteric Coated Aspirin 325mg | Apple Pectin + Aspirin | Placebo Comparator
Number analyzed (Participants) | 25 | 25 | 25 | 25
participants | 22 | 18 | 20 | 23

2. Primary Outcome: Time to Flushing
Description: The time it took, in minutes, for a participant to experience any flushing. Time to flush for individuals that did not experience flushing within 6 hours was set to 360 minutes.
Time Frame: 6 hours after dosing
Population: All participants randomized to the study completed the study. Each arm had 25 participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Apple-pectin 2000mg | Regular Non-enteric Coated Aspirin 325mg | Apple Pectin + Aspirin | Placebo Comparator
Number analyzed (Participants) | 25 | 25 | 25 | 25
minutes | 75.4 (51.7) | 48.7 (33.8) | 58.8 (42.5) | 58.1 (66.2)

3. Primary Outcome: Duration of Flushing
Description: The amount of time, in minutes, that flushing lasted. Duration of individuals without experience flushing within 6 hours was set to 0 minutes.
Time Frame: 6 hours after dosing
Population: All participants randomized to the study completed the study. Each arm had 25 participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Apple-pectin 2000mg | Regular Non-enteric Coated Aspirin 325mg | Apple Pectin + Aspirin | Placebo Comparator
Number analyzed (Participants) | 25 | 25 | 25 | 25
minutes | 43.3 (35.7) | 52.7 (53.5) | 58.3 (40.2) | 88 (66)

4. Primary Outcome: Maximum Flushing Severity Score
Description: Flushing assessment performed hourly for six hours. Assessment of severity done using the validated visual analog scale (VAS) flushing assessment tool (FAST). Severity rated using a VAS from mild (1-3), moderate (4-6), severe (7-9) to very severe (10). The maximum severity score was the maximum severity score of each individual during the 6 hours of monitoring time period.
Time Frame: 6 hours after dosing
Population: All participants randomized to the study completed the study. Each arm had 25 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apple-pectin 2000mg | Regular Non-enteric Coated Aspirin 325mg | Apple Pectin + Aspirin | Placebo Comparator
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale | 3.2 (2.7) | 2.8 (2.6) | 3.3 (2.5) | 3.6 (2.6)

ADVERSE EVENTS:
Arm/Group | Apple-pectin 2000mg | Regular Non-enteric Coated Aspirin 325mg | Apple Pectin + Aspirin | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Limitations include: pilot design, small sample size, short duration of a one-time niacin dose, utilization of only one niacin formulation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes